CLINICAL TRIAL: NCT01065649
Title: Effect of Nortriptyline in the Cortical Representation of Heartburn in Patients With Nonerosive Reflux Disease
Brief Title: Effect of Nortriptyline in Cortical Representation of Heartburn in Nonerosive Reflux Disease (NERD) Patients
Acronym: NORGERD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidade de Passo Fundo (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Fernando Fornari, PhD, Universidade de Passo Fundo
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 0102.0.398.000-09
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: reflux disease; heartburn
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn | interventions — Nortriptyline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nortriptyline (Experimental): 20 NERD patients will be treated with nortriptyline 10 mg a day in the first 7 days and 25 mg a day in the following 14 days
  Interventions: Drug: Nortriptyline
- Placebo (Placebo Comparator): Placebo arm
  Interventions: Drug: Nortriptyline; Drug: Placebo arm

INTERVENTIONS:
Drug: Nortriptyline — It will be administered per oral 10 mg a day in the first 7 days and then 25 mg a day in the last 14 days
Drug: Placebo arm — Placebo per oral for 21 days, equal to nortriptyline
  Arms: Placebo

SUMMARY:
Patients with nonerosive reflux disease (NERD) are less responsive to standard treatment with proton pump inhibitors. The hypothesis of this study was that nortriptyline in analgesic doses may decrease heartburn perception and its corresponding cortical activity measured by magnetic resonance image. Therefore, the aim of this study was to assess the cortical representation of heartburn in patients with NERD under treatment with nortriptyline and placebo.

ELIGIBILITY:
Inclusion Criteria:

* more than 17 years old, heartburn at least twice a week, naive to antireflux medications and antidepressive agents

Exclusion Criteria:

* active esophagitis at endoscopy, contraindications to nortriptyline use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Cortical representation of heartburn | 3 months

SECONDARY OUTCOMES:
Subjective assessment of heartburn | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Kozma, Passo Fundo, Rio Grande do Sul, Brazil